## **COVER PAGE**

## STATISTICAL ANALYSIS PLAN

OFFICIAL TITLE: The Correlation Between The Hopelessness Level and Self-Care

Agency In Patients Receiving Hemodialysis Treatment

DATE OF DOCUMENT: November 20, 2020

## Statistical Analysis Plan

The data were analyzed and assessed in computer environment through SPSS 22 program. Descriptive statistics for variables were given as number, percentages, arithmetic mean, and standard deviation. The compliance of the data to normal distribution was tested with the Shapiro Wilk test. Mann Whitney-U Test was used in the comparison of two groups and Kruskal Wallis Test was used in the comparison of more than two groups. The correlation between the study variables was evaluated with Spearman's Correlation analysis. The statistical significance of the difference was accepted as p<0.05.